CLINICAL TRIAL: NCT06811857
Title: An Exploration of Hyperbaric Oxygen in the Treatment of Flap Ischaemic Necrosis After Breast Cancer Surgery
Brief Title: This Study Aims to Explore the Efficacy of Hyperbaric Oxygen in the Treatment of Flap Ischaemic Necrosis After Breast Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1048-03
Record Dates: First submitted 2025-01-21; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Flap Necrosis; Flap Ischemia
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyperbaric oxygen group (Experimental): The hyperbaric group is given a total of 30-40 sessions of hyperbaric oxygen therapy (100% oxygen at a pressure of 2.0 ATA) and povidone-iodine wet compresses.
  Interventions: Device: hyperbaric oxygen therapy and povidone-iodine wet compresses
- Normal group (Active Comparator): The control group is given wet compresses of povidone-iodine.
  Interventions: Other: wet compresses of povidone-iodine

INTERVENTIONS:
Device: hyperbaric oxygen therapy and povidone-iodine wet compresses — The hyperbaric oxygen group receives 30-40 sessions of hyperbaric oxygen therapy (100% oxygen at a pressure of 2.0 ATA) and povidone-iodine wet compresses.
  Arms: hyperbaric oxygen group
Other: wet compresses of povidone-iodine — wet compresses of povidone-iodine
  Arms: Normal group

SUMMARY:
The expectation of our study was to explore the efficacy of using hyperbaric oxygen to rescue flap ischaemic necrosis after breast cancer surgery.

DETAILED DESCRIPTION:
Hyperbaric oxygen is commonly used to improve tissue oxygen saturation rescue flap ischemia, and treatment of diabetic foot ulcers. In the current study, there are also a number of case reports attempting to explore the role of hyperbaric oxygen in the treatment of postoperative skin flaps and nipple areola necrosis after breast surgery and significant efficacy has been obtained. Our study expects to use the treatment of hyperbaric oxygen to save patients with signs of flap ischemic necrosis after breast cancer surgery and to improve the quality of life and prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. understand the study procedure, participate in the study voluntarily and sign the informed consent form
2. aged ≥ 18 years and ≤ 60 years, female
3. ECOG 0-2
4. patients with The SKIN Score Degree of B-D and The SKIN area of 1-3 in the Clavien-Dindo classification after breast cancer surgery；

Exclusion Criteria:

1. Contraindications to hyperbaric oxygen therapy: lung disease (severe chronic obstructive airway disease, herpetic lung disease, acute or chronic lung infection, uncontrolled asthma, untreated pneumothorax), history of previous middle ear surgery, middle ear disease (Eustachian tube dysfunction, recurrent episodes of vertigo), eye disease (retinal detachment).
2. Pregnancy or lactation.
3. any other condition that the investigators think the patient is unsuitable for participation in the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The SKIN Area Score of Clavien-Dindo classification | At baseline, weekly during HBO treatment (up to 8 weeks), 2 weeks after the end of HBO treatment, 4 weeks after the end of HBO treatment

SECONDARY OUTCOMES:
NAC necrosis Degree | At baseline, weekly during HBO treatment (up to 8 weeks), 2 weeks after the end of HBO treatment, 4 weeks after the end of HBO treatment
Number of times for hyperbaric oxygen treatment | at the end of the study (at 3 month)
Interval between surgery and hyperbaric oxygen treatment | baseline
Breast-Q questionnaire | At baseline, end of hyperbaric oxygen treatment(at 6-8 weeks), 2 weeks after end of hyperbaric oxygen treatment, 4 weeks after end of hyperbaric oxygen treatment
  The BREAST-Q is a rigorously developed patient-reported outcome measure (PROM) designed to evaluate outcomes among women undergoing different types of breast surgery from the patient perspective.
side effects of hyperbaric oxygen treatment | During hyperbaric oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang Kun Wang, PhD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol